CLINICAL TRIAL: NCT03872323
Title: Comparison Between Open and Endovascular Surgical Techniques to Manage Vascular Injuries
Brief Title: Open and Endovascular Surgical Treatment for Artery Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinan Military General Hospital (Other)
Responsible Party: Principal Investigator, Li Min, Vice Director, Jinan Military General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 960HP20190045
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Artery Injury
Keywords: Artery Injury; Surgery; Endovascular Repair; Peripheral Arteries
MeSH Terms: interventions — Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular treatment (Active Comparator)
  Interventions: Procedure: Endovascular treatment
- Open surgery (Active Comparator)
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: Endovascular treatment — The arteries injuries are repaired by endovascular treatment.
  Arms: Endovascular treatment
Procedure: Open surgery — The arteries injuries are repaired by open surgical operation.
  Arms: Open surgery

SUMMARY:
Traumatic injuries of peripheral arteries are often associated with multiple injuries, massive hemorrhage, state of shock, and loss of blood supply, as well as with high mortality. Traditionally, an open surgical approach is suggested for the management of artery injury. With the advancement of endovascular techniques, the traditional open vascular exposure and vessel repair are no longer the only option available. The purpose of this study is to compare the effectiveness, long-term safety and explore the safety and efficacy factors between open and endovascular surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

Injuries in the peripheral arteries; Loss of blood supply to the remote area; High-risk emergency artery reconstruction; Participate in the study voluntarily, accept follow up study. -

Exclusion Criteria:

Bleeding can be easily control; There is contraindications for surgical operation. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
5-year treatment success rate | 60 months
  Treatment success is defined as restored blood flow without clinical complications.

SECONDARY OUTCOMES:
Technically success rate of surgery | immediately after surgery
Surgery-related complications or death | 60 months
Currence of stenosis of target lesion | 60 months
Device-related serious adverse events | 60 months
Target lesion was treated by interventional or surgical therapy once again | 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- 960 Hospital of PLA, Jinan, Shandong, China